CLINICAL TRIAL: NCT01315457
Title: Asian Multinational Retrospective Analysis for Infectious Complications in Patients Treated With Alemtuzumab
Brief Title: Infections Associated With the Use of Alemtuzumab
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: National Taiwan University Hospital (Other); Dr Cipto Mangunkusumo General Hospital (Other); Asan Medical Center (Other); Soon Chun Hyang University (Other); Chonnam National University (Other); Chonbuk National University (Other); Chulalongkorn University (Other); Queen Mary Hospital, Hong Kong (Other); Yonsei University (Other); Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Won Seog Kim, Professor, Samsung Medical Center
Other Study IDs: 2009-03-006
Record Dates: First submitted 2011-03-13; First posted 2011-03-15 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Patients Treated With Alemtuzumab
Keywords: alemtuzumab, infection, prophylaxis, treatment
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Alemtuzumab: Patients treated with alemtuzumab

SUMMARY:
The aim of this study is to propose infection prophylaxis from Asian multinational retrospective analysis of infectious complications in patients who were treated with alemtuzumab

ELIGIBILITY:
Inclusion Criteria:

* Patients received alemtuzumab as a treatment for hematologic malignancy ex. non-Hodgkin lymphoma Acute myeloid leukemia Aplastic anemia

Exclusion Criteria:

* Patients did not receive alemtuzumab

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients received alemtuzumab as a treatment for hematologic malignancy
Sampling Method: Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2009-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Infectious event | one year
  Any infectious complication occurred within one year after the use of alemtuzumab

CONTACTS AND LOCATIONS:
Overall Officials: Won Seog Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (5):
- Queen Mary Hospital, Hong Kong, China
- Cipto Mangunkusumo General Hospital, Jakarta, Indonesia
- Samsung Medical Center, Seoul, South Korea
- National Taiwan University Hospital, Teipei, Taiwan
- Chulalongkorn University, Bangkok, Thailand